CLINICAL TRIAL: NCT06168656
Title: Investigating the Effects of Mobile Application for Expectant Fathers About Preparation for Birth and Parenthood on Fear of Childbirth and Paternal Attachment
Brief Title: Examining a Mobile App's Impact on Expectant Fathers' Fear of Childbirth and Paternal Attachment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Busra Degirmenciler, Lecturer, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-60116787-020-301336
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Mobile Application; Expectant Fathers; Antenatal Education
Keywords: Mobile application; Antenatal Education; Fatherhood; Mobile Health

STUDY DESIGN:
Intervention Model Description: Single blind pre-post test randomized controlled design
Who Masked: Participant
Masking Description: Single
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The experimental group will use a mobile application intervention developed for expectant fathers.
  Interventions: Behavioral: Mobile Application
- No Intervention (No Intervention): Control group receive routine care.

INTERVENTIONS:
Behavioral: Mobile Application — The mobile application will include the following features:
  Direct Message Section: This section will allow expectant fathers to ask specialized questions directly to experts or specialists.
  Forum Section: Expectant fathers can use this section to engage in discussions and connect with each other.
  Education Section: This section is specifically designed to cater to the educational needs of expectant fathers.
  Arms: Experimental

SUMMARY:
Historically, reproduction and childbirth have conventionally been seen solely as a transition into motherhood and as matters primarily concerning the women. Expectant fathers often experience fear and stress in the perinatal period. Gender roles dictate that men should exude strength and self-assuredness. Hence, it leads expectant fathers to withhold their fears and emotions. Expectant fathers seek specific information about the process and may struggle with emotional expression. Fathers who overlook their own needs are unable to provide adequate support to their partners. Consequently, expectant mothers are more prone to experiencing heightened levels of stress, anxiety, and depression, and they may lean towards opting for cesarean deliveries. Additionally, they might persist in engaging in risky behaviors, such as smoking, and face challenges in maintaining breastfeeding. Support provided to expectant fathers leads to a positive influence on the health of both mothers and newborns. The development of technology has led to significant increase in the utilization of mobile devices within the healthcare. The implementation of mobile device interventions does not increase the workload on institutions and healthcare professionals. Hence, it can be utilized to address the needs of expectant fathers. For this reason, the aim of this study is to develop a mobile application to reduce expectant fathers' fear of childbirth and enhance paternal attachment.

DETAILED DESCRIPTION:
This study was planned as a parallel, single-blind, pre-post-test randomized controlled experimental study in which two groups (experiment-control) will be compared. The block randomization method will be used. The expectant fathers who will participate in the research will be reached through social media networks related to parenthood (Facebook and Instagram accounts) and the data will be collected from expectant fathers who are suitable for the sample characteristics through mobile application. The sample size was calculated in the G*power statistics program by utilizing the data of a study in which on expectant parents using a mobile application intervention was previously performed (α =0.05, d=0.80). Accordingly, it was found that 16 expectant fathers should be taken for each group to sampling for 80% power. Considering that there might be losses, the number of samples was increased by 40% and it was planned to include a total of 54 expectant fathers in the study. Intention-to-treat analysis will be performed to manage bias and losses. A pilot application will be conducted for 4 weeks with 6 expectant fathers regarding the usability of the mobile application and these expectant fathers will not be included in the study. At the end of 4 weeks, feedback will be received from the expectant fathers participating in the pilot application with the mobile application evaluation form. Necessary changes will be made in the mobile application in line with the feedback.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and above,
* Users of smartphones and social media,
* Willing to participate in the research,
* Proficient in understanding, speaking, and writing in Turkish,
* At least completed primary education,
* First-time fathers,
* Have not attended any antenatal education program,
* Have internet access and have used any mobile application before,
* Spouses with low-risk pregnancies in the 20-28 weeks gestational age and without a cesarean indication will be eligible for participation.

Exclusion Criteria:

* Fathers who have previously experienced childbirth before the post-test.
* Fathers who wish to withdraw from the research.
* Fathers who do not complete the educational program will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Expectant Fathers
Enrollment: 54 (Estimated)
Dates: Start 2023-12-31 (Estimated); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Fear of Birth Scale (FOBS) | Baseline and 6 weeks after
  This scale was developed by Haines et al. in 2011 to measure the fear of childbirth. In the scale, the participants were asked to rate their feelings by marking the statements (a) 'calm/worried' (b) 'no fear/strong fear' on two 100 mm lines to answer the question "How do you feel right now about the approaching birth?". Cronbach's Alpha internal consistency coefficient of the scale was 0.91. The cut-off score of the scale was 50. Participants who obtained a score of 50 or above were considered to fear of childbirth.
Paternal Antenatal Attachment Scale-PAAS | Baseline and 6 weeks after
  The PAAS was developed by Condon in 1993. The scale comprises 16 items. Each item of the scale focuses on measuring the father's emotions, attitudes, behaviors, and thoughts toward the developing fetus during pregnancy, with most items based on fathers' experiences in the last two weeks. Items are rated on a five-point Likert scale ranging from 1 to 5, with a total score range of 16-80. Lower scores indicate less antenatal attachment.
Introductory Information Form | Baseline
  This form includes sociodemographic questions such as age, gestational week, education level, employment status, and economic situation.
Mobile Application Evaluation Form | 4 weeks after the pilot intervention.
  This researcher-designed form assesses user satisfaction with the mobile app, gathering feedback on usability and content following the pilot application.